CLINICAL TRIAL: NCT03665246
Title: Evaluation of the iMBC/ECD Model on Maternal Mental Health and Child Development in Ghana
Brief Title: Evaluation of the iMBC/ECD Model in Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Catholic Relief Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-0020
Record Dates: First submitted 2018-08-20; First posted 2018-09-11 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Early Childhood Development
Keywords: ECD; maternal mental health; early childhood development; Ghana; ASQ; SRQ20; Integrated Mothers and Babies Course; maternal and child health

STUDY DESIGN:
Intervention Model Description: The present study is a cluster randomized trial (CRT) of 32 program groups with 16 groups randomly assigned to receive the intervention program (iMBC/ECD + C-PrES) and 16 groups randomly assigned to receive the control program (C-PrES only).The main reason for including randomization is to reduce the risk of selection bias. The unit of inference for this CRT is at the individual level but the unit of randomization is the C-PrES group (cluster) level due to issues of program feasibility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (iMBC/ECD + C-PrES) (Experimental): The intervention group of women/children dyads who consent will receive 14 sessions of the Integrated Mothers and Babies Course/Early Childhood Development (iMBC/ECD) curriculum in addition to the C-PrES curriculum. Upon completion of 14 sessions, women will continue to receive MNCHN and ECD messages and group-based iMBC booster sessions every 3 months.
  Interventions: Behavioral: Integrated Mothers and Babies Course
- Control (C-PrES) (No Intervention): The control group of women/children dyads who consent will have exposure to 14 sessions of the C-PrES curriculum which promotes the adoption of key MNCHN behaviors (e.g. newborn care, exclusive breastfeeding, etc.). Upon completion of 14 sessions, women will continue to receive MNCHN and ECD messages.

INTERVENTIONS:
Behavioral: Integrated Mothers and Babies Course — The Integrated Mothers and Babies Course/Early Childhood Development (iMBC/ECD) will be implemented along side normal C-PrES programming (key MNCHN behaviors). The iMBC curriculum is a prevention model based on cognitive behavioral therapy with the aim of supporting pregnant women and mothers with children under two years of age to become more resilient, decrease risk for future depression, and manage daily stressors effectively. In addition, the updated version of the iMBC is integrated with selected early childhood development (ECD) messages. The integration of these messages is intended to increase mothers' knowledge of the stressors associated with pregnancy and parenting young children and promote early stimulation behaviors and bonding to support child development.
  Arms: Intervention (iMBC/ECD + C-PrES)

SUMMARY:
The Duke research team will work with Catholic Relief Services (CRS) and lead the design and implementation of a cluster-randomized trial in Northern Ghana to assess the impact of the Integrated Mothers and Babies Course & Early Childhood Development (iMBC/ECD) intervention on the mental wellbeing of mothers of children under 2 and their children's attainment of age-appropriate developmental milestones.

DETAILED DESCRIPTION:
Maternal psychological disorders around the time of pregnancy and childbirth have been identified as a key risk factor for poor child development outcomes in growth, cognition, and overall child health in low- and middle-income countries (LMICs). Maternal depression during a child's infancy predicts negative behavior and lower achievement scores, as well as increased absences in elementary school), and has been identified as a significant risk factor for poor infant growth in the developing world. There is considerable evidence to suggest that a community-based intervention, delivered by trained community volunteers, can have a significant impact on perinatal depression and child development outcomes. This cluster-randomized trial in Northern Ghana will assess the impact of the Integrated Mothers and Babies Course & Early Childhood Development (iMBC/ECD) intervention on the mental wellbeing of mothers of children under 2 and their children's attainment of age-appropriate developmental milestones. In Ghana, the iMBC/ECD will be implemented in the context of the Rural Emergency Health Service and Transport project (REST II). A key activity of REST II is Community Pregnancy Surveillance and Targeted Education Sessions (C-PrES). Routine C-PrES is delivered via educational group sessions that promote the adoption of key Maternal, Neonatal and Child Health and Nutrition (MNCHN) behaviors (e.g. newborn care, exclusive breastfeeding, etc.) among pregnant women and mothers of children under age two.

ELIGIBILITY:
Inclusion Criteria (Mother):

* 16 years or older
* Currently pregnant
* Attends C-PrES groups at the time of the baseline survey (West Mamprusi and Nabdam District)
* Plan to maintain residence in the community for at least 6 months
* Agrees to voluntary participation

(The participation of the child falls under the mother's consent. Once born, the child will be followed along with its mother as long as the mother continues participation in the study.)

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Age-appropriate Social-Emotional Development of Children Under 2 Years | 6 months post-intervention
  The Ages and Stages Questionnaire:Social Emotional-2 (ASQ: SE-2) will be used to assess the attainment of age-appropriate social emotional development. The questionnaire that is administered is based on the child's age in completed months:
  * ASQ:SE 2 Month Questionnaire: 1 month 0 days - 2 months 30 days
  * ASQ:SE 6 Month Questionnaire: 3 month 0 days - 8 months 30 days
  * ASQ:SE 12 Month Questionnaire: 9 months 0 days - 14 months 30 days
  * ASQ:SE 18 Month Questionnaire: 15 months 0 days - 20 months 30 days
  * ASQ:SE 24 Month Questionnaire: 21 months 0 days - 26 months 30 days
Maternal Depression/Anxiety | 6 months post-intervention
  The 9 item Patient Health Questionnaire (PHQ-9) will be used to asses the mental health (depression) of mothers of children under 2. The PHQ-9 score ranges from 0-27, with higher numbers indicating higher levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Joy Noel Baumgartner, PhD, Principal Investigator — Duke University
Locations (1):
- Catholic Relief Services, Tamale, Ghana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao J, Gallis JA, Ali M, Lillie M, Abubakr-Bibilazu S, Adam H, McEwan E, Awoonor-Williams JK, Hembling J, Baumgartner JN. The impact of a maternal mental health intervention on intimate partner violence in Northern Ghana and the mediating roles of social support and couple communication: secondary analysis of a cluster randomized controlled trial. BMC Public Health. 2021 Nov 4;21(1):2010. doi: 10.1186/s12889-021-12121-9. PMID 34736452
- [Derived] Mackness J, Gallis JA, Owusu RK, Ali M, Abubakr-Bibilazu S, Adam H, Aborigo R, Awoonor-Williams JK, Lillie M, McEwan E, Hembling J, Vasudevan L, Baumgartner JN. Prevalence and correlates of maternal early stimulation behaviors during pregnancy in northern Ghana: a cross-sectional survey. BMC Pregnancy Childbirth. 2021 Jan 4;21(1):4. doi: 10.1186/s12884-020-03476-9. PMID 33397319